CLINICAL TRIAL: NCT02789826
Title: Laparoscopic Versus Open Resection of Cancer Stomach Randomized Controlled Trial
Brief Title: Laparoscopic Versus Open Resection of Cancer Stomach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Ameen Taher, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU4958
Record Dates: First submitted 2016-05-22; First posted 2016-06-03 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Laparoscopic gastric cancer resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Patients allocated to the 'laparoscopic Gastrectomy' group will undergo laparoscopic gastrectomy. If, during surgery, laparoscopic resection does not seem feasible, the procedure may be converted to an open one.
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): Patients allocated to the 'Open Gastrectomy' group will receive gastrectomy via laparotomy. This group is considered the control group
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — Patients allocated to the 'laparoscopic gastrectomy' arm will receive gastrectomy via laparoscopy.
  Other Names: Minimally invasive gastrectomy
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — patients allocated to the 'Open gastrectomy' group will receive gastrectomy via laparotomy
  Arms: Open gastrectomy

SUMMARY:
The aim of surgical procedures for resection of cancer stomach is to resection of the tumor mass with safety margin and its drainage lymph nodes (lymphadenectomy).

There are two main types of techniques (open & laparoscopic) Many studies were done comparing these two techniques showed that Laparoscopic resection is superior in early postoperative recovery (less pain ,less bleeding and shorter hospital stay) but less radical than open resection (less safety margin & less lymphadenectomy) but because of the ongoing advances on laparoscopic surgery these results needs more and more revision.

So the investigators conduct this randomized controlled trial aiming at comparing open and laparoscopic resection of cancer stomach to choose the best surgical procedure for resection of cancer stomach.

DETAILED DESCRIPTION:
The surgical procedure for resection of cancer stomach aiming at resection of the tumor mass with safety margin and its drainage lymph nodes (lymphadenectomy).

# Tumor resection;

Will be done by one of the following techniques:

1. laparoscopic gastrectomy (totally laparoscopic, laparoscopy-assisted, and hand-assisted) types of gastrectomy (according to site of tumour)
2. Open gastrectomy (according to the site of tumor). # Lymphadenectomy; Will be done according to Japanese Gastric Cancer Association guidelines for optimal lymph node dissection levels for Early Gastric Cancer (1):

   * D1+alpha -(perigastric lymph node dissection) for mucosal cancer, for which EMR is not indicated and for histologically differentiated submucosal cancer of < 1.5 cm in diameter;
   * D1+ beta for preoperatively diagnosed submucosal cancer without lymph node metastasis (N0), for which D1+ alpha is not indicated, and for early cancer < 2.0 cm in diameter with only perigastric lymph node metastasis (N1);
   * D2 for early cancer > 2.0 cm in diameter. Follow up: all patients will be followed up clinically for the outcomes for each surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary carcinoma of the stomach, where the tumor is considered surgically resectable (T1-3, N0-1, M0).

Exclusion Criteria:

* Pregnancy.
* Infiltration to the( pancreas ,liver ,colon or vital vascular structure).
* Metastasis to the (liver, lung, brain, paraaortic LN involvement).
* Peritoneal deposit.
* Surgically unfit patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The number of lymph nodes in the postoperative spicement. | two weeks
  considered a prognostic factor for disease-free postoperative survival The more the number of lymph nodes the more radicality of the procesure

SECONDARY OUTCOMES:
Mortality | 30 days post-operative
  Measured as 30-day mortality rate
Postoperative complications | Postoperatively with follow-up to one year
  Complications will be graded according to the Clavien-Dindo classification, which grades complications with regard to necessary treatment for this complication. Also Long-term complications, such as hernia cicatricialis will be monitored
Peri-operative blood loss | during surgery, 1 day
  Laparoscopic gastrectomy is associated with less peri-operative blood loss. Blood loss will be measured in milliliters and compared to the conventional 'open' group.
Duration of Surgery | Peri-operatively, 1 day
  UsuallyLaparoscopic gastrectomy takes longer time to complete. The duration of the procedure will be registered in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A Hamad, Prof., Study Director — Assiut University- Faculty of Medicine; Mostafa M Sayed, Study Director — Assiut University- Faculty of Medicine; Mohamed G Taher, Principal Investigator — Assiut University- Faculty of Medicine- General surgery department
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No